CLINICAL TRIAL: NCT03707041
Title: A Single Centre, Randomised, Double-blind, Placebo-controlled, Phase Ib Study to Evaluate the Safety, Tolerability and Chemoprotective Antimalarial Activity of P218 Against Controlled Human Malaria Infection With Plasmodium Falciparum Sporozoite Challenge in Non-immune Healthy Adult Volunteers
Brief Title: Safety, Tolerability and Chemoprotective Activity of P218 in PfSPZ Challenge Model
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: SGS Life Sciences, a division of SGS Belgium NV (Other); Institute of Tropical Medicine, Belgium (Other); Washington University School of Medicine (Other); Swiss BioQuant (Industry); PrimeVigilance Ltd., UK (Industry); Biologic LLP, UK (Industry); Sanaria Inc. (Industry); FGK Representative Service B.V., The Netherlands (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMV_P218_17_01; 2018-003004-39 (EudraCT Number)
Record Dates: First submitted 2018-10-09; First posted 2018-10-16 (Actual); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Malaria
Keywords: malaria; PfSPZ Challenge; chemoprotection
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: In each of the three treatment cohorts, subjects will be randomly allocated to receive either P218 or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo capsules matched to the drug product with regard to appearance and taste
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- P218 1000 mg (Oral Capsules) - Cohort 1 (Experimental): Two administrations of 1000 mg P218 (capsules p.o.), 48 hours apart
  Interventions: Drug: P218 (1000 mg) Oral Capsules
- P218 Placebo Oral Capsules - Cohort 1 (Placebo Comparator): Two administrations of P218 placebo (capsules p.o.), 48 hours apart
  Interventions: Drug: Placebo Oral Capsules
- P218 1000 mg (Oral Capsules) - Cohort 2 (Experimental): One administration of 1000 mg P218 (capsules p.o.), 2 hours after PfSPZ Challenge and one administration of 1000 mg P218 (capsules p.o.), 48 hours after first administration.
  Interventions: Drug: P218 (1000 mg) Oral Capsules; Biological: PfSPZ Challenge
- P218 Placebo Oral Capsules - Cohort 2 (Placebo Comparator): One administration of P218 placebo (capsules p.o.), 2 hours after PfSPZ Challenge and one administration of P218 placebo (capsules p.o.,) 48 hours after first administration.
  Interventions: Drug: Placebo Oral Capsules; Biological: PfSPZ Challenge
- P218 100 mg (Oral Capsules) - Cohort 3 (Experimental): One administration of 100 mg P218 (capsules p.o.), 2 hours after PfSPZ Challenge and one administration of 100 mg P218 (capsules p.o.), 48 hours after first administration.
  Interventions: Drug: P218 (100 mg) Oral Capsules; Biological: PfSPZ Challenge
- P218 Placebo Oral Capsule - Cohort 3 (Active Comparator): One administration of P218 placebo (capsules p.o.), 2 hours after PfSPZ Challenge and one administration of P218 placebo (capsules p.o.), 48 hours after first administration.
  Interventions: Drug: Placebo Oral Capsules; Biological: PfSPZ Challenge

INTERVENTIONS:
Drug: P218 (1000 mg) Oral Capsules — 1000 mg P218 (4 x 250 mg capsules)
  Arms: P218 1000 mg (Oral Capsules) - Cohort 1; P218 1000 mg (Oral Capsules) - Cohort 2
Drug: Placebo Oral Capsules — Placebo capsules matched to the P218 capsules with regard to appearance and taste
  Arms: P218 Placebo Oral Capsule - Cohort 3; P218 Placebo Oral Capsules - Cohort 1; P218 Placebo Oral Capsules - Cohort 2
Drug: P218 (100 mg) Oral Capsules — 100 mg P218 (2 x 50 mg capsules)
  Arms: P218 100 mg (Oral Capsules) - Cohort 3
Biological: PfSPZ Challenge — 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)
  Arms: P218 100 mg (Oral Capsules) - Cohort 3; P218 1000 mg (Oral Capsules) - Cohort 2; P218 Placebo Oral Capsule - Cohort 3; P218 Placebo Oral Capsules - Cohort 2

SUMMARY:
This was a single centre, randomised, double-blind, placebo-controlled Phase Ib study, to evaluate the safety, tolerability and chemoprotective activity of P218 in a controlled P. falciparum sporozoite infection model.

Healthy men and women, aged 18 to 45 years were to be enrolled in 3 study cohorts and to be administered either P218 or placebo twice, 48 hours apart. Subjects in cohorts 2 and 3 were to be inoculated with P. falciparum sporozoites. Enrolment in cohorts was to proceed sequentially, to facilitate review of data by a Safety Review Team (SRT) before proceeding with a subsequent cohort.

In cohort 1, safety and tolerability of P218 was assessed. In cohorts 2 and 3, chemoprotective activity of P218 against malaria infection was assessed, as well as the Influence of time of initiation of the P218 treatment on the protective effect.

DETAILED DESCRIPTION:
This was a single centre, randomised, double-blind, placebo-controlled Phase Ib study, to evaluate the safety, tolerability and chemoprotective activity of P218 in a controlled P. falciparum sporozoite infection model.

32 healthy men and women, aged 18 to 45 years were to be enrolled in 3 cohorts of respectively 8, 12 and 12 subjects. A subject could be enrolled in one cohort only and was to be randomised in a 3:1 ratio, to receive two consecutive administrations, 48 hours apart, of either P218 or placebo. Enrolment in cohorts proceeded sequentially, to facilitate review of data by a Safety Review Team (SRT) before populating a subsequent cohort.

Cohort 1 consisted of 2 subgroups of subjects, to be enrolled sequentially: subgroup 1 was to be composed of 2 subjects: one to receive two 1000 mg doses of P218 and one to receive placebo twice. Subgroup 2 was to be composed of 6 subjects: five to receive two 1000 mg doses of P218 and one to receive placebo twice. Subjects in subgroup 2 would not be treated until 24 hours after second IMP administration in the last subject of subgroup 1 and only after review of the safety data from subgroup 1 by the PI. Duration of each subject treatment and follow-up in Cohort 1 was 9 days. Progression to Cohort 2 was subject to review of the safety and tolerability data by a SRT.

Cohort 2 consisted of three subgroups of subjects, to be enrolled sequentially. Subgroup 1 was to be composed of 2 subjects: one to receive two 1000 mg doses of P218 and one to receive placebo twice. Subgroups 2 and 3 were to be composed of 5 subjects each: four to receive two 1000 mg doses of P218 and one to receive placebo twice. Subjects in subgroup 2 would not be treated until 24 hours after second IMP administration in the last subject of subgroup 1. On Day 1, each subject in Cohort 2 would be administered 3200 P. falciparum sporozoites (PfSPZ Challenge) by direct venous inoculation (DVI). First administration of 1000 mg of P218 or placebo will take place 2 hours after PfSPZ Challenge DVI; second administration of 1000 mg of P218 or placebo would take place 48 hours later. As of Day 7, parasitemia in every subject was to be assessed daily until the installation of malarial infection or until Day 28. Overall duration of each subject observation in Cohort 2 was 35 days. Progression to Cohort 3 was subject to assessment of safety and parasitemia data, as well as malaria signs and symptoms by a SRT.

Cohort 3 was to consist of two subgroups each with 6 subjects, to be enrolled sequentially. Treatment was to be allocated in a ratio of 3 active: 1 placebo. In each subgroup, at least 1 subject was to receive placebo and the remaining subjects would receive two 100 mg doses of P218 48 hours apart. Subjects in subgroup 2 would not be inoculated until 24 hours after second IMP administration in the last subject of subgroup 1. On Day 1, subjects were to be administered 3200 P. falciparum sporozoites by DVI. As of Day 7, parasitemia in every subject was to be assessed daily until the installation of malarial infection or until Day 28. Overall duration of each subject observation in Cohort 3 is 35 days.

All subjects in Cohorts 2 and 3 would receive antimalarial rescue therapy, either upon installation of malarial infection or on Day 28 or if leaving the study prematurely.

In Cohort 1, safety and tolerability of two 1000 mg doses of P218 administered 48 hours apart was to be assessed over 9 days of observation. Pharmacokinetic assessments of P218 and its main metabolites were to take place over 9 days of observation.

In Cohorts 2 and 3, chemoprotective activity of two doses P218 (1000 mg or 100 mg respectively) administered 48 hours apart, were to be assessed over 28 days. Safety and tolerability of two doses of P218 (1000 mg or 100 mg respectively) administered 48 hours apart were to be assessed over 35 days of observation. Pharmacokinetic assessments of P218 would take place over 9 days of observation.

ELIGIBILITY:
Subjects meeting all of the following criteria are eligible to participate in this study:

1. Informed Consent Form signed voluntarily before any study-related procedure is performed, indicating that the subject understands the purpose of and procedures required for the study and is willing to participate in the study, including administration of rescue treatment.
2. Male or female, between 18 and 45 years old (extremes included) at screening.
3. Body weight of at least 50 kg and a body mass index (BMI) of 19 to 30 kg/m2 (extremes included).
4. Good general health without clinically relevant medical illness, physical exam findings including vital signs, and laboratory abnormalities as determined by the investigator.
5. Willing to adhere to the prohibitions and restrictions (see Section 4.3) specified in this protocol, including willingness to stay confined to the inpatient unit for required duration and willingness to avoid to travel outside of Benelux during the study period.
6. Female subjects should fulfil one of the following criteria:

   1. At least 1 year post-menopausal (amenorrhea >12 months and follicle-stimulating hormone (FSH) >30 mIU/mL) prior to screening;
   2. Surgically sterile (bilateral oophorectomy, hysterectomy or tubal ligation);
   3. Will use contraceptives as outlined in inclusion criteria 7 and 8.
7. Female subjects of childbearing potential must agree to the use of a highly effective method of birth control from screening visit to until 40 days after the last dose of IMP (covering a full menstrual cycle of 30 days starting after 5 half-lives of last dose of IMP).

   Note: Highly effective birth control methods include: combined (estrogen and progestogen containing) oral/intravaginal/transdermal hormonal contraception associated with inhibition of ovulation, progestogen-only oral/injectable/implantable hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner or sexual abstinence.
8. Male subjects who are sexually active with a female partner of childbearing potential must agree to the use of an effective method of birth control from the day of the first IMP dose until 100 days thereafter (covering a full sperm cycle of 90 days starting after 5 half-lives of last dose of IMP).

   Note: Medically acceptable methods of contraception that may be used by the subject and/or partner include sterilization and vasectomy or a double barrier option combining oral contraceptive, contraceptive vaginal ring, contraceptive injection, intrauterine device or etonogestrel implant.
9. Female subject has a negative pregnancy test at screening and upon admission in the clinical unit.

   Note: Pregnancy testing will consist of a serum β-human chorionic gonadotropin (β-HCG) test at screening and urine β-HCG tests at other visits, in all women.

   Inclusion Criteria - CHMI (controlled human malaria infection) specific:
10. Different ways of being reachable 24/7 (e.g. by mobile phone, regular phone or electronic mail) during the whole study period.

Subjects meeting any of the following criteria are excluded from participation in this study:

1. Nursing (lactating) women.
2. Participation in any other clinical drug or vaccine study within 30 days (or five half-lives for drugs) preceding the first dose of IMP (whichever is longer), or plans to participate in other investigational drug or vaccine research during the study period.
3. Blood product donation to any blood bank during the 8 weeks (whole blood) or 4 weeks (plasma and platelets) prior to admission in the clinical unit.
4. ECG outside normal range and deemed clinically relevant by the investigator. Examples of clinically significant ECG abnormalities for this study include:

   1. PR-interval >220 ms;
   2. QRS-complex >120 ms;
   3. QT interval corrected according to Bazett's formula (QTcB) or QT interval corrected according to Fridericia's formula [3] (QTcF) >450 ms;
   4. Pathologic Q wave;
   5. Significant ST-T wave changes;
   6. Left or right ventricular hypertrophy;
   7. Non-sinus rhythm except isolated premature atrial contractions and ventricular extrasystole <2 per 10 s ECG lead;
   8. Incomplete left bundle branch block, or complete or intermittent right or left bundle branch block;
   9. Second or third degree A-V heart block.
5. Seropositive human immunodeficiency virus (HIV) (antibody and antigen), hepatitis B virus (HBV) (hepatitis B surface antigen [HBsAg]) or hepatitis C virus (HCV) (antibody) tests.
6. History or presence of diagnosed food or known drug allergies (including but not limited to allergy to any of the antimalarial rescue medications to be used in the study, see Section 5.2), or history of anaphylaxis or other severe allergic reactions.

   Note: Subjects with seasonal allergies/hay fever, house dust mite or allergy to animals that are untreated and asymptomatic at the time of dosing can be enrolled in the study.
7. History of convulsion or severe head trauma.

   Note: A medical history of a single febrile convulsion during childhood is not an exclusion criteria.
8. History of serious psychiatric condition that may affect participation in the study or preclude compliance with the protocol, including but not limited to past or present psychoses, disorders requiring lithium, a history of attempted or planned suicide, more than one previous episode of major depression, any previous single episode of major depression lasting for or requiring treatment for more than 6 months, or any episode of major depression during the 5 years preceding screening.

   Note: The Beck Depression Inventory (Attachment 2) will be used as an objective tool for the assessment of depression at screening. In addition to the conditions listed above, subjects with a score of 20 or more on the Beck Depression Inventory and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) will not be eligible for participation. Subjects with a Beck score of 17 to 19 may be enrolled at the discretion of the Investigator if they do not have a history of the psychiatric conditions mentioned in this criterion and their mental state is not considered to pose additional risk to the health of the volunteer or to the execution of the study and interpretation of the data gathered.
9. A medical, occupational or family problem as a result of alcohol or illicit drug abuse during the past 12 months or current alcohol or illicit drug abuse or addiction (positive alcohol breath test or positive drug screen for amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine or opiates at screening or upon check-in at the clinical unit).

   Note: Excessive use of alcohol is an intake of >21 units per week for males and >14 units per week for females where one alcohol unit is defined as 10 mL or 8 g of pure alcohol. A single unit is equal to one 25-mL (single) measure of whisky (alcohol by volume [ABV] 40%), or a third of a pint of beer (190 mL; ABV 5-6%) or half a standard (175 mL) glass of wine (ABV 12%).
10. Subjects are non-smokers or ex-smokers for more than 90 days prior to screening or smoke no more than 5 cigarettes per day. If users of nicotine products (i.e. spray, patch, e-cigarette, etc.) they should use the equivalent of no more than 5 cigarettes per day. Subjects must agree to abstain from smoking while in the unit.
11. Use of any prescription drugs, herbal supplements (e.g. St John's Wort) or over-the-counter medication within 7 days or five half-lives (whichever is longer) prior to the first IMP administration, or an anticipated requirement for the use of these during the course of the study (See Section 6.2).

    Note: If necessary, the incidental use of non-steroidal anti-inflammatory drugs (NSAIDs), paracetamol (2g/day, 10 gr/week), vitamins and topical treatments may be acceptable after approval by the study Sponsor and will be documented in the eSource system. The use of nutritional supplements during this time that are not believed to have the potential to affect subject safety nor the overall results of the study, may be permitted on a case-by-case basis following approval by the Sponsor in consultation with the Investigator.
12. Any surgical or medical condition possibly affecting drug absorption (e.g. cholecystectomy, gastrectomy, bowel disease), distribution, metabolism or excretion.
13. Any history of gallbladder disease, including cholecystitis and/or cholelithiasis.
14. History of megaloblastic anaemia or folate deficiency.
15. Personnel (e.g. investigator, sub-investigator, research assistant, pharmacist, study coordinator or anyone mentioned in the delegation log) directly involved in the conduct of the study.
16. Any condition that in the opinion of the investigator would jeopardize the safety or rights of a person participating in the trial or would render the person unable to comply with the protocol.

    Exclusion Criteria - CHMI specific:
17. Glucose-6-phosphate dehydrogenase (G6PD) deficiency (due to possible hemolysis induced by primaquine treatment at study end in G6PD deficient subjects).
18. Personal history of malaria.
19. Volunteer has travelled to or lived in a malaria-endemic area for more than 4 weeks during the 12 months prior to first IMP administration, or spent any time in an endemic area during the 4 weeks prior to first IMP administration.
20. Plans to travel to malaria-endemic region during the study period up to last follow-up visit.
21. Previous participation in any malaria vaccine or CHMI study.
22. Falling in moderate or higher risk category for a fatal or non-fatal cardiovascular event within 10 years (≥5%) determined by a validated risk estimation system e.g. SCORE [13].
23. Use of medications known to interact with atovaquone-proguanil (Malarone®), artemether-lumefantrine (Riamet®) or primaquine (Primaquine®) such as cimetidine, metoclopramide or antacids, or an anticipated requirement for the use of these at any point during the study period (see Section 6.2).
24. Use of systemic antibiotics with known antimalarial activity within 30 days (or 5 half-lives whichever is longer) of first IMP administration (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones or azithromycin) or an anticipated requirement for the use of these during the study period (see Section 6.2).
25. Receipt of blood or blood-derived products (including immunoglobulin) within 3 months prior to screening. Receipt of packed red blood cells given for an emergent indication in an otherwise healthy person, and not required as ongoing treatment is not exclusionary (for example packed red blood cells emergently given during an elective surgery).

Note: In case of an out-of-range clinical laboratory test, vital sign or ECG value that will determine a subject's eligibility, or in case of a positive drug screen, a retest or expert evaluation can be requested. Results of any retest must be available prior to inoculation. The result of the retest will be considered for subject eligibility at the investigator's discretion. Subjects can be rescreened at the discretion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Donini, PhD, Study Director — MMV; Pieter-Jan Berghmans, MD, Principal Investigator — SGS Belgium NV
Locations (1):
- SGS Belgium NV Clinical Pharmacology Unit, Antwerp, Belgium

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the SGS Life Sciences Clinical Pharmacology Unit in Antwerp.
Pre-assignment Details: 61 subjects were screened, 32 subjects were enrolled and randomised.
Period: Overall Study
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 1 | P218 Placebo Oral Capsules - Cohort 1 | P218 1000 mg (Oral Capsules) - Cohort 2 | P218 Placebo Oral Capsules - Cohort 2 | P218 100 mg (Oral Capsules) - Cohort 3 | P218 Placebo Oral Capsule - Cohort 3
Started | 6 | 2 | 9 | 3 | 9 | 3
Completed | 6 | 2 | 9 | 3 | 9 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- P218 Placebo Oral Capsule - Cohorts 2 and 3: One administration of P218 placebo (capsules p.o.), 2 hours after PfSPZ Challenge and one administration of P218 placebo (capsules p.o.), 48 hours after first administration.
  Placebo Oral Capsules: Placebo capsules matched to the P218 capsules with regard to appearance and taste
  PfSPZ Challenge: 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)
- Total: Total of all reporting groups
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 1 | P218 Placebo Oral Capsules - Cohort 1 | P218 1000 mg (Oral Capsules) - Cohort 2 | P218 100 mg (Oral Capsules) - Cohort 3 | P218 Placebo Oral Capsule - Cohorts 2 and 3 | Total
Number analyzed (Participants) | 6 | 2 | 9 | 9 | 6 | 32
Age, Continuous [Median (Full Range); unit: years] | 33.5 [24 to 45] | 24.5 [24 to 25] | 36.0 [22 to 40] | 35.0 [23 to 42] | 34.5 [33 to 42] | 29.5 [22 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4 | 4 | 0 | 12
  Male | 3 | 1 | 5 | 5 | 6 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 2 | 9 | 7 | 6 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 6 | 2 | 9 | 9 | 6 | 32

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Number of TEAEs
Description: Incidence, severity and relationship to the treatment of observed or self-reported treatment emergent adverse events (TEAEs) after two single doses of 1000 mg P218 administered 48 hours apart in healthy adult volunteers.
Time Frame: 9 days
Measure: Count of Participants; unit: Participants
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 1 | P218 Placebo Oral Capsules - Cohort 1
Number analyzed (Participants) | 6 | 2
Participants
  Subjects with any TEAE | 2 | 1
  Subjects without any TEAE | 4 | 1

2. Primary Outcome: Cohorts 2 and 3: Geometric Mean Time From PfSPZ Challenge to First Quantitative Polymerase Chain Reaction (qPCR) Outcome Equal or Greater Than 250 Asexual Parasites Per mL of Blood
Description: Chemoprotective activity of two single doses of 1000 mg P218 administered 2 hours after PfSPZ Challenge and 48 hours later in healthy adult volunteers
Time Frame: Number of days from PfSPZ Challenge DVI to positive parasitaemia, or 28 days
Measure: Geometric Mean (90% Confidence Interval); unit: Days
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 2 | P218 100 mg (Oral Capsules) - Cohort 3 | P218 Placebo Oral Capsule - Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 6
Days | 28.000 [28.000 to 28.000] | 25.822 [22.396 to 29.771] | 10.615 [9.918 to 11.360]

3. Secondary Outcome: Cohorts 2 and 3: Number of P218 TEAEs
Description: Incidence, severity and relationship to the P218 treatment of observed or self-reported treatment emergent adverse events in non-immune healthy adult volunteers after two single doses of 1000 mg P218 administered 48 hours apart in a controlled human malaria infection (PfSPZ Challenge)
Time Frame: 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 2 | P218 100 mg (Oral Capsules) - Cohort 3 | P218 Placebo Oral Capsule - Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 6
Participants
  Any P218-related TEAEs | 1 | 0 | 0
  No P218-related TEAEs | 8 | 9 | 6

4. Secondary Outcome: Cohorts 2 and 3: Number of PfSPZ Challenge TEAEs
Description: Incidence, severity and relationship to the PfSPZ Challenge of observed or self-reported treatment emergent adverse events in non-immune healthy adult volunteers before and after P218 administration
Time Frame: 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 2 | P218 100 mg (Oral Capsules) - Cohort 3 | P218 Placebo Oral Capsule - Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 6
Participants
  Subjects with any TEAE | 9 | 1 | 6
  Subjects without any TEAE | 0 | 8 | 0

5. Secondary Outcome: Cohorts 2 and 3: Malaria Clinical Score at the Time of Introduction of Rescue Therapy
Description: The malaria clinical score consists of 14 signs/symptoms frequently associated with malaria and graded using a 4-point scale (absent: 0; mild: 1; moderate: 2; severe: 3) and summed to generate a total malaria clinical score (maximum score possible is 42): headache, myalgia (muscle ache), arthralgia (joint ache), fatigue/lethargy, malaise (general discomfort/uneasiness), chills/shivering/rigors, sweating/hot spells, anorexia, nausea, vomiting, abdominal discomfort, fever, tachycardia and hypotension.
  To determine severity of the 14 signs/symptoms the CTCAE grading scale grade 1 - 5 was used. Mild (1) equates to CTCAE grade 1, Moderate (2) equates to CTCAE grade 2 and Severe (3) equates to CTCAE grade 3 or above. Individual scores for each symptom as well as the total score were recorded.
Time Frame: On the day of positive parasitaemia or on Day 28
Measure: Median (Full Range); unit: Malaria Clinical Score
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 2 | P218 100 mg (Oral Capsules) - Cohort 3 | P218 Placebo Oral Capsule - Cohorts 2 and 3
Number analyzed (Participants) | 9 | 9 | 6
Malaria Clinical Score | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 1.00 [0.0 to 5.0]

6. Secondary Outcome: Cohorts 1, 2 and 3: P218 AUC[0-48h] - Day 1
Description: Area under the P218 plasma concentration-time curve from first administration to 48 hours after first administration
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 1 | P218 1000 mg (Oral Capsules) - Cohort 2 | P218 100 mg (Oral Capsules) - Cohort 3
Number analyzed (Participants) | 6 | 9 | 9
h*ng/mL | 16752 (6958) | 13865 (2663) | 1296 (332)

7. Secondary Outcome: Cohort 1: P218-beta-acyl-glucuronide-OH AUC[48-96h]
Description: Area under the P218-beta-acyl-glucuronide-OH plasma concentration-time curve from 48 hours after first P218 administration to 96 hours after first P218 administration
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- P218 1000 mg - Cohort 1: Two administrations of 1000 mg P218 (capsules p.o.), 48 hours apart
  P218 (1000 mg) Oral Capsules: 1000 mg P218 (4 x 250 mg capsules)
Arm/Group | P218 1000 mg - Cohort 1
Number analyzed (Participants) | 6
h*ng/mL | 27283 (7106)

8. Secondary Outcome: Cohorts 1, 2 and 3: P218 Cmax - Day 1
Description: Maximum observed P218 plasma concentration after each P218 administration
Time Frame: 9 days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 1 | P218 1000 mg (Oral Capsules) - Cohort 2 | P218 100 mg (Oral Capsules) - Cohort 3
Number analyzed (Participants) | 6 | 9 | 9
ng/mL | 7482 (3889) | 7241 (2983) | 856 (338)

9. Secondary Outcome: Cohorts 1, 2 and 3: P218 Tmax - Day 1
Description: Time to P218 Cmax after each P218 administration
Time Frame: 9 days
Measure: Median (Full Range); unit: hours
Arm/Group | P218 1000 mg (Oral Capsules) - Cohort 1 | P218 1000 mg (Oral Capsules) - Cohort 2 | P218 100 mg (Oral Capsules) - Cohort 3
Number analyzed (Participants) | 6 | 9 | 9
hours | 1.00 [1.00 to 4.00] | 1.00 [0.55 to 1.50] | 1.00 [0.50 to 2.00]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of informed consent until the last study-related activity for each subject. A maximum period of 37 days for cohort 1, and 63 days for cohorts 2 and 3.
Groups:
- P218 Placebo - Cohort 1: Two administrations of P218 placebo (capsules p.o.), 48 hours apart
  Placebo Oral Capsules: Placebo capsules matched to the P218 capsules with regard to appearance and taste
- P218 1000 mg - Challenge - Cohort 2: One administration of 1000 mg P218 (capsules p.o.), 2 hours after PfSPZ Challenge and one administration of 1000 mg P218 (capsules p.o.), 48 hours after first administration.
  P218 (1000 mg) Oral Capsules: 1000 mg P218 (4 x 250 mg capsules)
  PfSPZ Challenge: 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)
- P218 100 mg - Challenge - Cohort 3: One administration of 100 mg P218 (capsules p.o.), 2 hours after PfSPZ Challenge and one administration of 100 mg P218 (capsules p.o.), 48 hours after first administration.
  P218 (100 mg) Oral Capsules: 100 mg P218 (2 x 50 mg capsules)
  PfSPZ Challenge: 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)
- P218 Placebo - Challenge - Cohorts 2 and 3: One administration of P218 placebo (capsules p.o.), 2 hours after PfSPZ Challenge and one administration of P218 placebo (capsules p.o.), 48 hours after first administration.
  Placebo Oral Capsules: Placebo capsules matched to the P218 capsules with regard to appearance and taste
  PfSPZ Challenge: 3200 P. falciparum Sporozoites by direct venous inoculation (DVI)
Arm/Group | P218 1000 mg - Cohort 1 | P218 Placebo - Cohort 1 | P218 1000 mg - Challenge - Cohort 2 | P218 100 mg - Challenge - Cohort 3 | P218 Placebo - Challenge - Cohorts 2 and 3
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/2 | 0/9 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/2 | 0/9 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 1/2 | 9/9 | 1/9 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P218 1000 mg - Cohort 1 (N=6) | P218 Placebo - Cohort 1 (N=2) | P218 1000 mg - Challenge - Cohort 2 (N=9) | P218 100 mg - Challenge - Cohort 3 (N=9) | P218 Placebo - Challenge - Cohorts 2 and 3 (N=6)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza-like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel Puncture Site Haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lip Dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03707041/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT03707041/SAP_001.pdf